CLINICAL TRIAL: NCT02602925
Title: Tight Control Dose Reductions of Biologics in Psoriasis Patients With Low Disease Activity: A Randomized Pragmatic Trial
Brief Title: Tight Control Dose Reductions of Biologics in Psoriasis Patients With Low Disease Activity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONDOR
Record Dates: First submitted 2015-10-09; First posted 2015-11-11 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2016-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Randomized, controlled non-inferiority study
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose decrease (Experimental): Patients receive daily practice care, but doses of etanercept, adalimumab or ustekinumab will be lowered: intervals of drug-administration will be prolonged stepwise with tight control of disease activity and DLQI. First, the dose will be decreased to 66-70% of the normal dose (by interval prolongation with a factor 1.5). If patients remain in a state of low disease activity, the dose will be further reduced to 50% (by doubling the original interval). Each step will be analyzed after three months, or when the patient visits earlier due to complaints.
  Interventions: Other: Dose decrease
- Usual care (Other): Patients will continue treatment with the normal dose and treatment regimens will be based on usual daily practice care. Treatment decisions are made at the discretion of the treating physician.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Dose decrease — Treatment strategy change: dose decrease based on PASI and DLQI
  Arms: Dose decrease
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
Rationale/hypothesis: Moderate-to-severe psoriasis can be treated with biologics.

Objective To investigate whether the dose of biologics can be reduced in patients with psoriasis with stable disease.

Study design: A pragmatic, multicentre, randomized, controlled, non-inferiority study with cost-effectiveness analysis.

Study population: Patients with disease remission using normal dose of biologics.

Intervention: 120 patients will be randomized into two groups: (1) dose reduction and (2) normal dose.

Main study parameters/endpoints: The primary outcome is clinical effectiveness. Secondary outcomes are: health-related quality of life (HRQoL), number and time to disease flares, costs, health status, anti-drug antibody formation and serious adverse events

DETAILED DESCRIPTION:
Rationale/hypothesis: Moderate-to-severe psoriasis can be treated with biologics. These drugs have significantly improved the quality of life of psoriasis patients, but are very expensive drugs that should be used as efficiently as possible. In addition, the long-term safety profile can probably be improved if patients receive the lowest effective dose.

Objective To investigate whether the dose of biologics can be reduced in patients with psoriasis with stable disease: Is dose reduction non-inferior to the current practice regarding clinical effectiveness? Secondary aims are: to investigate what influence dose tapering has on quality of life, whether there are predictors for successful dose reduction, and to determine the cost-effectiveness of dose reduction.

Study design: A pragmatic, multicentre, randomized, controlled, non-inferiority study with cost-effectiveness analysis.

Study population: Patients who used a biologic for at least 6 months (etanercept, adalimumab, ustekinumab) can be included if they have long-term stable low disease activity. Low disease activity is defined as a PASI score (Psoriasis Area and Activity Score) <5 and a health-related quality of life score ≤5 (Dermatology Quality of life index: DLQI).

Intervention: 120 patients will be randomized into two groups: (1) dose reduction guided by PASI and DLQI (n=60, intervention) and (2) maintenance of normal dosage (n=60, usual care).

Main study parameters/endpoints: The primary outcome is clinical effectiveness. Secondary outcomes are: health-related quality of life (HRQoL), number and time to disease flares, costs, health status, anti-drug antibody formation and serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Sustained low disease activity as described above on the dose as advised by the label.
* Established diagnosis of plaque psoriasis.
* Receiving treatment with adalimumab, etanercept, or ustekinumab for at least 6 months.*
* Age ≥18 years.
* Ability to understand informed consent, read and answer questionnaires.

Exclusion Criteria:

* Psoriasis itself is not the main reason for biologic prescription (e.g. when a patient has RA and psoriasis, and RA is the main reason for the biologic).
* Concomitant use of immunosuppressants other than methotrexate or acitretin for psoriasis.
* Severe comorbidities with short life-expectancy (e.g. metastasized tumour).
* Presumed inability to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Disease-activity | 1 year
  Disease-activity measured by Psoriasis Area and Severity Index (PASI), effectiveness measure used in most psoriasis trials.

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL-DLQI) | 1 year
  HRQoL(Dermatology Life Quality Index (DLQI)
Number of patients with 1 or more persistent flares | 1 year
  Number of patients with 1 or more persistent flares (persistent flare is defined as at least 3 months PASI increase >5 or DLQI >5)
Disease-activity measured with HsCRP | 1 year
  High-sensitivity CRP, a possible marker for disease-activity
Predictors for succesful dose decrease (treatment and patient characteristics) | 1 year
  For both groups, patient (sex, age, PsA, comorbidities) and treatment characteristics (antibody formation, through levels of drug, dose of biologic, drug pauses, use of concomitant antipsoriatic systemic drugs (dose and duration of use), use of topical therapies during treatment (steroid class and duration of use)) will be collected. These will be used to identify predictors for successful dose reduction.
Anti-drug antibody levels against etanercept, adalimumab or ustekinumab | 1 year
  Anti-drug antibodies (AU/mL) of the used biologic (etanercept, adalimumab or ustekinumab) will be measured using enzyme-linked immunosorbent assay or ELISA. Measures will take place at baseline and every study visit (week 0, 12, 24, 36 and 49). Anti-drug antibody levels will be used to assess whether they predict successful dose decrease.
Drug trough levels of etanercept, adalimumab or ustekinumab | 1 year
  Drug trough levels (mg/l) of the used biologic (etanercept, adalimumab or ustekinumab) will be measured using enzyme-linked immunosorbent assay or ELISA. Measures will take place at baseline and every study visit (aprox. every 3 months). Anti-drug antibody levels will be used to assess whether they predict successful dose decrease.
Number of serious adverse events per patient | 1 year
  All serious adverse events (SAE) during study participation and their causal relation with the biologic will be assessed.
Costs related to medical consumption | 1 year
  For cost-effectiveness analyses, questionnaires iMTA MCQ (medical consumption questionnaire) will be administered in each group at every study visit except baseline (week 12, 24, 36, 49).Data will be incorporated and presented in a cost-effectiveness analysis.
Costs related to productivity | 1 year
  For cost-effectiveness analyses, questionnaire iMTA PCQ (productivity cost questionnaire) will be administered in each group at every study visit except baseline (week 12, 24, 36, 49).Data will be incorporated and presented in a cost-effectiveness analysis.
Health status (SF36) | 1 year
  SF-36v2 questionnaire will be used to measure health status. Outcomes will be presented seperataly (scores for mental and physical health domain); but will also be incorporated and presented in a cost-effectiveness analysis. Questionnaire will be administered every study visit except baseline (week 12, 24, 36, 49).

CONTACTS AND LOCATIONS:
Overall Officials: E de Jong, MD, Principal Investigator — Dept. of Dermatology, Radboudumc, The Netherlands
Locations (6):
- Netherlands (6):
  - ZGT hospital, Almelo
  - Gelre hospitals, Apeldoorn
  - Slingeland Hospital, Doetinchem
  - St. Anna hospital, Geldrop
  - ZGT, Hengelo
  - Radboudumc, dept of dermatology, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Atalay S, van den Reek JMPA, den Broeder AA, van Vugt LJ, Otero ME, Njoo MD, Mommers JM, Ossenkoppele PM, Koetsier MI, Berends MA, van de Kerkhof PCM, Groenewoud HMM, Kievit W, de Jong EMGJ. Comparison of Tightly Controlled Dose Reduction of Biologics With Usual Care for Patients With Psoriasis: A Randomized Clinical Trial. JAMA Dermatol. 2020 Apr 1;156(4):393-400. doi: 10.1001/jamadermatol.2019.4897. PMID 32049319
- [Derived] Atalay S, van den Reek JMPA, van Vugt LJ, Otero ME, van de Kerkhof PCM, den Broeder AA, Kievit W, de Jong EMGJ. Tight controlled dose reduction of biologics in psoriasis patients with low disease activity: a randomized pragmatic non-inferiority trial. BMC Dermatol. 2017 May 8;17(1):6. doi: 10.1186/s12895-017-0057-6. PMID 28482858